CLINICAL TRIAL: NCT00057642
Title: Improving Hispanic Retention in Antidepressant Therapy
Brief Title: Improving Retention of Hispanics Receiving Antidepressant Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #4358; R21MH066388 (NIH); DSIR SE-SC
Record Dates: First submitted 2003-04-04; First posted 2003-04-07 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2008-09

CONDITIONS: Depression; Depressive Disorder
Keywords: Hispanic Americans
MeSH Terms: conditions — Depression; Depressive Disorder | interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sertraline, venlafaxine, bupropion (Other): This is an open trial so there is only one arm using standard antidepressant medications.
  Interventions: Drug: Sertraline; Drug: Venlafaxine Extended Release

INTERVENTIONS:
Drug: Sertraline
Drug: Venlafaxine Extended Release

SUMMARY:
This study will develop an intervention that will increase the retention of Hispanics with major depression in antidepressant therapy.

DETAILED DESCRIPTION:
Despite major advances in the treatment of psychiatric disorders, Hispanics continue to underutilize mental health services relative to their own mental health needs. Cultural factors are important causes of underutilization. To date, however, attempts to boost utilization by improving the cultural congruence of psychiatric services have not focused on retaining Hispanics in antidepressant therapy.

Motivational Interviewing (MI) is a time-limited psychotherapy that has successfully improved treatment retention among patients with dually diagnosed substance abuse and psychiatric disorders. During Phase I of this study, MI is adapted for use as an adjunctive therapy with antidepressant treatment and culturally adapted to Hispanic participants. In Phase II, participants receive sertraline for 12 weeks and participate in four sessions of MI therapy as a supplementary intervention designed to encourage treatment retention. Participants who are intolerant to sertraline or have an inadequate response by Week 6 are switched to venlafaxine ER while continuing to receive MI and to complete study assessments. A follow-up interview is conducted 6 months after the termination of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic Statistical Manual, 4th edition criteria for Major Depressive Disorder
* Patients who self-identify as Hispanic and are Spanish-dominant, English-dominant, or bilingual
* Acceptable methods of contraception
* Hamilton Depression Rating Scale score >= 18 at Visit 1
* Sertraline or venlafaxine ER is clinically appropriate

Exclusion Criteria:

* History of schizophrenia, bipolar affective disorder, schizoaffective disorder, depression with psychotic symptoms, or organic brain syndrome
* DSM-IV criteria for alcohol or substance abuse or dependence during the 6 months prior to screening
* Pregnancy or breast-feeding
* At risk for committing suicide
* Clinically significant renal, pulmonary, cerebrovascular, cardiovascular, gastrointestinal, or endocrine disorders
* Glaucoma, history of increased intraocular pressure (IOP), or at risk for having increased IOP
* Untreated or unstable hypertension
* Clinically significant laboratory abnormalities or abnormal electrocardiogram
* Medical conditions that might interfere with the process of drug absorption, metabolism, or elimination
* Clinically significant thyroid dysfunction (except patients who are stable and asymptomatic on thyroid replacement therapy)
* Current or past history of seizure disorder (except febrile seizure in childhood)
* History of failed sertraline or venlafaxine treatment for at least 4 weeks at adequate doses
* Allergy or hypersensitivity to sertraline or venlafaxine
* History of two failed selective serotonin reuptake inhibitor (SSRI) trials for major depression at adequate doses and duration
* Monoamine oxidase inhibitors (MAOIs) or fluoxetine within 4 weeks prior to screening, or other SSRIs, antidepressants, neuroleptics, mood stabilizers, buspirone, benzodiazepines, or other psychotropic drugs (except zolpidem for insomnia) within 2 weeks prior to screening
* Electroconvulsive Therapy (ECT) within the last 3 months
* Effective medication or psychotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2002-09; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Retention percentage | 12 weeks
  The proportion of weeks in treatment

SECONDARY OUTCOMES:
Depressive symptoms on the Hamilton Depression scale | 12 weeks
Number of days in treatment | 84 days
  Sum of days in treatment
Functional impairment on the Sheehan Disability Scale | 12 weeks
Perceived quality of life | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Lewis-Fernandez, MD, Principal Investigator — Columbia University, NY State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Derived] Lewis-Fernandez R, Balan IC, Patel SR, Sanchez-Lacay JA, Alfonso C, Gorritz M, Blanco C, Schmidt A, Jiang H, Schneier F, Moyers TB. Impact of motivational pharmacotherapy on treatment retention among depressed Latinos. Psychiatry. 2013 Fall;76(3):210-22. doi: 10.1521/psyc.2013.76.3.210. PMID 23965261